CLINICAL TRIAL: NCT00482729
Title: A Randomized, Double-Blind, Active-Comparator Controlled, Clinical Trial to Study the Efficacy and Safety of MK0431A for the Treatment of Patients With Type 2 Diabetes Mellitus (T2DM)
Brief Title: MK0431A Comparative Study in Patients With Type 2 Diabetes (0431A-079)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431A-079; MK0431A-079; 2007_548
Record Dates: First submitted 2007-05-31; First posted 2007-06-05 (Estimated); Results first posted 2010-03-15 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Metformin; Sitagliptin Phosphate, Metformin Hydrochloride Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Arm 1: drug
  Interventions: Drug: sitagliptin phosphate (+) metformin hydrochloride
- 2 (Active Comparator): Arm 2: active comparator
  Interventions: Drug: metformin

INTERVENTIONS:
Drug: sitagliptin phosphate (+) metformin hydrochloride — sitagliptin/Metformin HCl 50/500 mg tablet bid, titrating up to sitagliptin/Metformin HCl 50/1000 mg tablet over 4 weeks; for a 44-wk treatment period.
  Other Names: MK0431A; Janumet™
  Arms: 1
Drug: metformin — metformin 500 mg tablet bid, titrating up to 1000 mg tablets bid for a 44-wk treatment period
  Arms: 2

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of an investigational treatment for type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Patient has type 2 diabetes mellitus
* Patient is greater than or equal to 18 and less than or equal to 78 years of age on the day of signing the consent
* Patient has Hb1Ac greater than or equal to 7.5% and is appropriate for oral therapy
* Patient has not been on any antihyperglycemic agent (AHA) in the last 4 months
* Patient is a male, or a female who is unlikely to conceive

Exclusion Criteria:

* Patient has type 1 diabetes mellitus or history of ketoacidosis

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1246 (Actual)
Dates: Start 2007-06-19 (Actual); Primary Completion 2008-11-03 (Actual); Study Completion 2009-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Reasner C, Olansky L, Seck TL, Williams-Herman DE, Chen M, Terranella L, Johnson-Levonas AO, Kaufman KD, Goldstein BJ. The effect of initial therapy with the fixed-dose combination of sitagliptin and metformin compared with metformin monotherapy in patients with type 2 diabetes mellitus. Diabetes Obes Metab. 2011 Jul;13(7):644-52. doi: 10.1111/j.1463-1326.2011.01390.x. PMID 21410627
- [Result] Olansky L, Reasner C, Seck TL, Williams-Herman DE, Chen M, Terranella L, Mehta A, Kaufman KD, Goldstein BJ. A treatment strategy implementing combination therapy with sitagliptin and metformin results in superior glycaemic control versus metformin monotherapy due to a low rate of addition of antihyperglycaemic agents. Diabetes Obes Metab. 2011 Sep;13(9):841-9. doi: 10.1111/j.1463-1326.2011.01416.x. PMID 21535346

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient In: 26-Jun-2007; Last Patient Last Visit for end of study: 28-Apr-2009; Two-hundred four medical clinics in the United States (US) and 5 in Puerto Rico.
Pre-assignment Details: Patients 18-78 years of age with type 2 diabetes mellitus (T2DM) with inadequate glycemic control (hemoglobin A1c [A1C] >7.5% at screening visit) who were appropriate for treatment with oral antihyperglycemic therapy and had not been on an anti-hyperglycemic agent (AHA) in the last 4 months were eligible to participate.
Groups:
- Sita/Met FDC: The Sitagliptin/Metformin Fixed Dose Combination (Sita/Met FDC) group includes data from patients randomized to receive treatment with oral tablets of Sita/Met initiated at a dose of 50/500 mg twice a day (b.i.d.) The dose was to have been up-titrated over 4 weeks to 50/1000 mg b.i.d.; however, patients could stay in the study on a minimum dose of Sita/Met 50/500 mg b.i.d. if a higher dose was not tolerated.
- Metformin: The Metformin group includes data from patients randomized to receive treatment with oral tablets of metformin initiated at a dose of 500 mg twice a day (b.i.d.) The dose was to have been up-titrated over 4 weeks to 1000 mg b.i.d. ; however, patients could stay in the study on a minimum dose of Sita/Met 50/500 mg b.i.d. if a higher dose was not tolerated.
Period: Overall Study
Arm/Group | Sita/Met FDC | Metformin
Started | 626 (Site 079011301 was identified as non-compliant and 1 patient was excluded from all analysis) | 624 (Site 079011301 was identified as non-compliant and 3 patients were excluded from all analysis)
Completed Phase A | 484 | 482
Completed Phase B | 409 | 406
Completed | 409 | 406
Not Completed | 217 | 218
Not completed — Adverse Event | 29 | 33
Not completed — Creatinine/Creatinine Clearance Criteria | 0 | 2
Not completed — Hyperglycemia Criteria | 7 | 5
Not completed — Lack of Efficacy | 4 | 16
Not completed — Lost to Follow-up | 86 | 66
Not completed — Physician Decision | 10 | 7
Not completed — Pregnancy | 4 | 2
Not completed — Protocol Violation | 10 | 18
Not completed — Withdrawal by Subject | 67 | 69

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sita/Met FDC | Metformin | Total
Number analyzed (Participants) | 625 | 621 | 1246
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (10.5) | 50.0 (10.5) | 49.7 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 272 | 266 | 538
  Male | 353 | 355 | 708
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 17 | 24 | 41
  Black | 82 | 88 | 170
  White | 508 | 489 | 997
  Other | 18 | 20 | 38
Hemoglobin A1c (A1C) [Mean (Standard Deviation); unit: Percent] | 9.91 (1.83) | 9.83 (1.77) | 9.87 (1.80)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (A1C) at Week 18
Description: A1C is measured as percent. Thus, this change from baseline reflects the Week 18 A1C percent minus the Week 0 A1C percent.
Time Frame: Baseline and Week 18
Population: The Full Analysis Set (FAS) included all patients who received at least 1 dose of double-blind study therapy, had a baseline value and ≥ 1 post-baseline value for this outcome. Data after initiation of additional AHA were treated as missing. For FAS with no data at Week 18, the last post-baseline observed measurement was carried forward to Week 18.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Sita/Met FDC | Metformin
Number analyzed (Participants) | 559 | 564
Percent | -2.37 [-2.49 to -2.24] | -1.76 [-1.88 to -1.64]
Statistical Analysis 1: Comparison: Sita/Met FDC vs Metformin; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment, baseline A1C; Mean Difference (Net) = -0.60, 95% CI [-0.78 to -0.43]

2. Secondary Outcome: Number of Patients With A1C < 7.0% at Week 18
Time Frame: Week 18
Population: The Full Analysis Set (FAS) included all patients who received at least 1 dose of double-blind study therapy, had a baseline value and ≥1 post-baseline value for this outcome. Data after initiation of additional AHA were treated as missing. For FAS with no data at Week 18, the last post-baseline observed measurement was carried forward to Week 18.
Measure: Number; unit: Participants
Arm/Group | Sita/Met FDC | Metformin
Number analyzed (Participants) | 559 | 564
Participants
  Patients with A1C <7.0% at Week 18 | 275 | 193
  Patients with A1C ≥7.0% at Week 18 | 284 | 371
Statistical Analysis 1: Comparison: Sita/Met FDC vs Metformin; Test type: Superiority or Other; p < 0.001, ANCOVA — Based on a test of the odds ratio = 1, comparing the odds of having A1C <7.0% at Week 18 in the Sita/Met FDC group vs. the Metformin group; Model terms: treatment, baseline A1C; Odds Ratio (OR) = 2.07, 95% CI [1.60 to 2.69] — This parameter estimate and 95% confidence interval correspond to the odds of having A1C <7.0% at Week 18 in the Sita/Met FDC group vs. the Metformin group

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 18
Description: FPG is measured as mg/dL. Thus, this change from baseline reflects the Week 18 FPG mg/dL minus the Week 0 FPG mg/dL.
Time Frame: Baseline and Week 18
Population: The Full Analysis Set (FAS) included all patients who received at least 1dose of double-blind study therapy, had a baseline value and ≥1 post-baseline value for this outcome. Data after initiation of additional AHA were treated as missing. For FAS with no data at Week 18, the last post-baseline observed measurement was carried forward to Week 18.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sita/Met FDC | Metformin
Number analyzed (Participants) | 560 | 566
mg/dL | -69.4 [-74.1 to -64.6] | -53.7 [-58.4 to -48.9]
Statistical Analysis 1: Comparison: Sita/Met FDC vs Metformin; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment, baseline A1C; Mean Difference (Net) = -15.7, 95% CI [-22.4 to -9.0]

4. Other Pre Specified Outcome: Change From Baseline in A1C at Week 44
Description: A1C is measured as percent. Thus, this change from baseline reflects the Week 44 A1C percent minus the Week 0 A1C percent.
Time Frame: Baseline and Week 44
Population: The Full Analysis Set (FAS) included all patients who received at least 1 dose of double-blind study therapy, had a baseline value and ≥1 post-baseline value for this outcome. Data after initiation of additional AHA were included. For FAS with no data at Week 44, the last post-baseline observed measurement was carried forward to Week 44.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Sita/Met FDC | Metformin
Number analyzed (Participants) | 560 | 569
Percent | -2.25 [-2.38 to -2.12] | -1.77 [-1.89 to -1.64]
Statistical Analysis 1: Comparison: Sita/Met FDC vs Metformin; Test type: Superiority or Other; Mean Difference (Net) = -0.48, 95% CI [-0.67 to -0.30] — This is a difference in least squares means, based on an ANCOVA model with terms for treatment and baseline (i.e., Week 0) A1C

5. Other Pre Specified Outcome: Number of Patients With A1C < 7.0% at Week 44
Time Frame: Week 44
Population: The Full Analysis Set (FAS) included all patients who received at least 1dose of double-blind study therapy, had a baseline value and ≥1 post-baseline value for this outcome. Data after initiation of additional AHA were included. For FAS with no data at Week 44, the last post-baseline observed measurement was carried forward to Week 44.
Measure: Number; unit: Participants
Arm/Group | Sita/Met FDC | Metformin
Number analyzed (Participants) | 560 | 569
Participants
  Patients with A1C <7.0% at Week 44 | 258 | 173
  Patients with A1C ≥7.0% at Week 44 | 302 | 396
Statistical Analysis 1: Comparison: Sita/Met FDC vs Metformin; Test type: Superiority or Other; Odds Ratio (OR) = 2.11, 95% CI [1.63 to 2.73] — This parameter estimate and 95% confidence interval correspond to the odds of having A1C <7.0% at Week 44 in the Sita/Met FDC group vs. the Metformin group, based on a logistic regression model with terms for treatment and baseline (i.e., Week 0) A1C

ADVERSE EVENTS:
Time Frame: Week 0 through Week 44
Description: 1 patient in the Sita/Met FDC group and 3 patients in the Metformin group from Site 079011301, which was identified as non-compliant with some of the requirements of Good Clinical Practice. For this reason, data from all four randomized patients at this site were deemed unreliable and were excluded from the primary efficacy and safety analysis.
Arm/Group | Sita/Met FDC | Metformin
Serious Adverse Events (participants affected / at risk) | 28/625 | 38/621
Other Adverse Events (participants affected / at risk) | 173/625 | 185/621
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sita/Met FDC (N=625) | Metformin (N=621)
Any Cardiac Disorders (Cardiac disorders) | 5 | 6
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 3
Myocardial infarction (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Any Gastrointestinal Disorders (Gastrointestinal disorders) | 2 | 2
Food poisoning (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1
Any General Disorders and Administration site Conditions (General disorders) | 1 | 3
Adverse drug reaction (General disorders) | 0 | 1
Electrocution (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 1
Any Hepatobiliary disorders (Hepatobiliary disorders) | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Any Infections and Infestations (Infections and infestations) | 6 | 6
Appendicitis (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 1
Hepatitis C (Infections and infestations) | 0 | 1
Pneumonia streptococcal (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Any Injury, Poisoning and Procedural Complications (Injury, poisoning and procedural complications) | 2 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 1
Skull fractured base (Injury, poisoning and procedural complications) | 0 | 1
Any Metabolism and Nutrition Disorders (Metabolism and nutrition disorders) | 1 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Diabetic foot (Metabolism and nutrition disorders) | 1 | 1
Any Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 5
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Any Nervous System Disorders (Nervous system disorders) | 1 | 5
Carotid artery disease (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Transient ischaemic attack (Nervous system disorders) | 1 | 2
Any Pregnancy, puerperium and perinatal conditions (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Any Psychiatric Disorders (Psychiatric disorders) | 2 | 3
Anxiety (Psychiatric disorders) | 1 | 0
Panic attack (Psychiatric disorders) | 1 | 0
Schizophrenia (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 2
Any Renal and Urinary Disorders (Renal and urinary disorders) | 2 | 2
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Neurogenic bladder (Renal and urinary disorders) | 0 | 1
Postrenal failure (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Any Respiratory, Thoracic and Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Any Vascular Disorders (Vascular disorders) | 2 | 4
Aneurysm (Vascular disorders) | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 1
Aortic stenosis (Vascular disorders) | 1 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sita/Met FDC (N=625) | Metformin (N=621)
Any Gastrointestinal Disorders (Gastrointestinal disorders) | 107 | 136
Diarrhoea (Gastrointestinal disorders) | 86 | 112
Nausea (Gastrointestinal disorders) | 37 | 44
Any Infections and infestations (Infections and infestations) | 62 | 57
Nasopharyngitis (Infections and infestations) | 33 | 26
Upper respiratory tract infection (Infections and infestations) | 30 | 31
Any Nervous system disorders (Nervous system disorders) | 35 | 23
Headache (Nervous system disorders) | 35 | 23

LIMITATIONS AND CAVEATS:
Site 079011301 was non-compliant with Good Clinical Practice (GCP). Data from the 4 patients at this site are included in the Participant Flow summary, but are excluded from all other summaries and analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.